CLINICAL TRIAL: NCT04773756
Title: Evaluation of Sofosbuvir and Daclatasvir Combo in COIVD-19 Patients in Egypt (Single Center Study)
Brief Title: Evaluation of Sofosbuvir and Daclatasvir Combo in COIVD-19 Patients in Egypt
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Amr Aly Abd Elmoety, Professor, Internal Medicine Department, Alexandria University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0305032
Record Dates: First submitted 2021-02-22; First posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Covid19
Keywords: Sofosbuvir; Daclatasvir
MeSH Terms: conditions — COVID-19 | interventions — Sofosbuvir; daclatasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sofosbuvir / Daclatsvir (Other): A drug used in the treatment of HCV infection, given in the same dose 400mg and 60 mg respectively once daily for 14 days
  Interventions: Drug: Sofosbuvir 400 MG/ Daclatasvir 60mg

INTERVENTIONS:
Drug: Sofosbuvir 400 MG/ Daclatasvir 60mg — Giving these two drugs for treatment of COVID patients

SUMMARY:
Sofosbuvir has been recently recommended as a possible antiviral for COVID-19, based on structural studies and multiple alignment analysis. By comparing the positive-stranded RNA genomes of HCV and SARS-CoV-2, it has been postulated that sofosbuvir might be an optimal nucleotide analogue to repurpose for COVID-19 treatment

ELIGIBILITY:
Inclusion Criteria:

* mild- moderate COVID-19 confirmed by PCR

Exclusion Criteria:

1. Patients on renal dialysis
2. Severe COVID-19 cases
3. Patients on amiodarone therapy (given the reported FDA warning of an interaction between amiodarone and sofosbuvir that might lead to severe bradycardia).
4. Children < 12 years
5. Pregnant and breast feeding women
6. Exacerbation of hepatitis B

Ages: 12 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-12 (Actual)

PRIMARY OUTCOMES:
evaluate the combined effect of Sofosbuvir and Daclatasvir in treatment of patients with mild-moderate Covid-19. | it is estimated to be 2 weeks
  The study assesses the incidence of resolution of symptoms in COVID patients after taking Sofosbuvir and Daclatasvir for 14 days by doing PCR and the result to be negative

CONTACTS AND LOCATIONS:
Overall Officials: Amr Abd elmoety, PhD, Principal Investigator — Alexandria University, Faculty of Medicine
Locations (1):
- Amr Aly Abd elmoety, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No